CLINICAL TRIAL: NCT02708680
Title: A Randomized, Placebo-controlled, Double-blind, Multicenter Phase 2 Study of Atezolizumab With or Without Entinostat in Patients With Advanced Triple Negative Breast Cancer, With a Phase 1b Lead in Phase
Brief Title: Randomized Phase 2 Study of Atezolizumab and Entinostat in Patients With aTN Breast Cancer With Phase 1b Lead In
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Syndax Pharmaceuticals (Industry)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNDX-275-0602
Record Dates: First submitted 2016-03-09; First posted 2016-03-15 (Estimated); Results first posted 2023-09-14 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — entinostat; atezolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Entinostat plus Atezolizumab (Active Comparator): Participants in this arm will receive entinostat in combination with atezolizumab.
  Phase 1b Dose Determination: The initial 3 to 6 participants will receive entinostat at a starting dose of 5 milligrams (mg) (Dose Group 1) on Days 1, 8, and 15 along with atezolizumab 1200 mg via intravenous (IV) infusion on Day 1 of each 21-day cycle. If the 5 mg dose exceeds the maximum tolerated dose (MTD), then a 3 mg dose of entinostat (Dose Group -1) will be evaluated in the same manner. If the -1 dose level exceeds the MTD, then a 2 mg dose of entinostat (Dose Group -2) will be evaluated.
  Phase 2 Dose Expansion: Participants will receive the RP2D identified in the Dose Determination Phase.
  Interventions: Drug: Entinostat; Drug: Atezolizumab
- Placebo plus Atezolizumab (Placebo Comparator): Participants in this arm will receive placebo in combination with atezolizumab 1200 mg.
  Interventions: Drug: Atezolizumab; Drug: Placebo

INTERVENTIONS:
Drug: Entinostat — An orally available histone deacetylases inhibitor (HDAC).
  Other Names: SNDX-275; MS-275
  Arms: Entinostat plus Atezolizumab
Drug: Atezolizumab — A humanized, engineered monoclonal antibody of IgG1 isotype against the protein programmed cell death ligand 1 (PD-L1).
  Other Names: MPDL3280A
Drug: Placebo — A pill containing no active drug ingredient
  Arms: Placebo plus Atezolizumab

SUMMARY:
The purpose of this study is to determine the safety and tolerability of entinostat used in combination with atezolizumab in participants with Advanced Triple Negative Breast Cancer (aTNBC). Additionally, the purpose of the study is to assess how effective entinostat and atezolizumab are in combination in participants with aTNBC.

DETAILED DESCRIPTION:
SNDX-275-0602 is a Phase 1b/2 study evaluating the combination of entinostat plus atezolizumab in participants with aTNBC. The study has 2 phases: an open-label Dose Determination Phase (Phase 1b) followed by an Expansion Phase (Phase 2). The Expansion Phase will evaluate the efficacy and safety of entinostat when administered at the RP2D with atezolizumab in participants with aTNBC in a randomized, double-blind, placebo-controlled setting.

Safety will be assessed during the study by documentation of AEs, clinical laboratory tests, physical examinations, vital sign measurements, electrocardiograms (ECGs), and Eastern Cooperative Oncology Group (ECOG) performance status. Adverse events of special interest (AESI) will be collected and reviewed in a manner consistent with serious adverse event reporting procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Has histologically or cytologically confirmed triple negative breast carcinoma that is either metastatic (stage IV of the TNM classification) or locally recurrent and not amenable to local curative treatment.
2. Evidence of measurable, locally recurrent or metastatic disease based on imaging studies within 28 days before the first dose of study drug.
3. Has received at least 1, but no more than 2, prior lines of systemic therapy for locally recurrent and/or metastatic disease.
4. If participant has a history of treated asymptomatic CNS metastases they are eligible, provided they meet all of the following criteria: participant has measurable disease outside CNS; participant does not have metastases to midbrain, pons, medulla or spinal cord; participant is not on corticosteroids as therapy for CNS disease (anticonvulsants at a stable dose are allowed); participant has not had whole-brain radiation within 6 weeks prior to study enrollment; participant has stable CNS disease as demonstrated by at least 4 weeks of stability between the last intervention scan and the study screening scan.
5. ECOG performance status of 0 or 1.
6. Has acceptable, applicable laboratory parameters.
7. Female participants must not be pregnant; willing to use 2 methods of birth control/abstinence if applicable through 120 days after the last dose of study drug.
8. Experienced resolution of toxic effect(s) of the most recent prior anti-cancer therapy to Grade <1 (except alopecia or neuropathy).
9. Able to understand and give written informed consent and comply with study procedures.

Exclusion Criteria:

1. Diagnosis of immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
2. Active autoimmune disease including active diverticulitis, symptomatic peptic ulcer disease, colitis, or inflammatory bowel disease that has required systemic treatment in past 2 years.
3. Previously treated with a PD-1/PD-L1-blocking antibody or a histone deacetylase inhibitor.
4. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating Investigator, including, but not limited to: history of immune deficiencies or autoimmune disease; myocardial infarction or arterial thromboembolic events within 6 months prior to screening or severe or unstable angina, New York Heart Association (NYHA) Class III or IV disease, or a QTc interval > 470 msec; uncontrolled hypertension or diabetes mellitus; another known malignancy that is progressing or requires active treatment; active infection requiring systemic therapy; known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
5. Any contraindication to oral agents or significant nausea and vomiting, malabsorption, or significant small bowel resection that, in the opinion of the investigator, would preclude adequate absorption.
6. Received a live vaccine within 30 days of the first dose of treatment.
7. Prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to enrollment or who has not recovered from AEs due to mAb agents administered more than 4 weeks earlier.
8. Prior chemotherapy within 3 weeks, targeted small molecule therapy or radiation therapy within 2 weeks prior to enrollment, or who has not recovered (i.e., ≤Grade 1 at enrollment) from AEs due to a previously administered agent.
9. Received transfusion of blood products or administration of colony stimulating factors within 4 weeks prior to the first dose of treatment.
10. Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of study drug.
11. Currently receiving treatment with any other agent listed on the prohibited medication list.
12. If female, is pregnant, breastfeeding, or expecting to conceive starting with the screening visit through 120 days after the last dose of study drug.
13. Known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies).
14. Known active hepatitis B or hepatitis C.
15. Allergy to benzamide or inactive components of entinostat.
16. History of allergies to any active or inactive ingredients of atezolizumab.
17. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Slamon, MD, Principal Investigator — University of California, Los Angeles
Locations (29):
- United States (19):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - CBCC Global Research at Comprehensive Blood and Cancer Center, Bakersfield, California
  - St. Jude Medical Center, Fullerton, California
  - Los Angeles Hematology Oncology Medical Group, Glendale, California
  - Torrance Memorial Cancer Care Associates, Redondo Beach, California
  - SLO Oncology and Hematology Health Center, San Luis Obispo, California
  - Central Coast Medical Oncology Group, Santa Maria, California
  - UCLA Hematology/Oncology - Santa Monica, Santa Monica, California
  - Saint Mary's Regional Cancer Center, Grand Junction, Colorado
  - Office of Human Research, Hollywood, Florida
  - Orlando Health, Inc., Orlando, Florida
  - Ft. Wayne Hematology and Oncology, Fort Wayne, Indiana
  - Ft. Wayne Medical Oncology & Hematology, Inc, Fort Wayne, Indiana
  - Cancer Center of Kansas, Wichita, Kansas
  - Frauenshuh Cancer Center at Park Nicollet Health Service, Saint Louis Park, Minnesota
  - Saint Barnabas Medical Cancer Center, Livingston, New Jersey
  - Hope Women's Cancer Centers, Asheville, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
- Georgia (10):
  - Cancer Center of Adjara Autonomous Republic, Batumi, Adjara
  - Saint Nikolozi Surgery and Oncological Centre, Kutaisi, Imereti
  - Unimed Adjara - Oncology Center, Kutaisi, Imereti
  - Health House, Tbilisi
  - Institute of Clinical Oncology, Tbilisi
  - New Vision University Hospital, Tbilisi
  - Cancer Research Center, Tbilisi
  - S. Khechinashvili, University Hospital, Tbilisi
  - Multiprofile Clinic Consilium Medulla, Tbilisi
  - Research Institute of Clinical Medicine, Tbilisi

IPD SHARING:
Plan to Share IPD: No
An independent data safety monitoring board (DSMB) will be established for the Phase 2 portion of this study to act in an advisory capacity to the Sponsor with respect to safeguarding the interests of trial patients and assessing the safety of the interventions administered during the trial.

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1b Dose Determination: Entinostat Plus Atezolizumab.; Phase 2 Expansion Phase: Entinostat Plus Atezolizumab: Participants received entinostat 5 mg in combination with atezolizumab 1200 mg.
- Phase 2 Expansion Phase: Placebo Plus Atezolizumab: Participants received placebo in combination with atezolizumab 1200 mg.
Period: Overall Study
Arm/Group | Phase 1b Dose Determination: Entinostat Plus Atezolizumab. | Phase 2 Expansion Phase: Entinostat Plus Atezolizumab | Phase 2 Expansion Phase: Placebo Plus Atezolizumab
Started | 8 | 40 | 41
Received At Least 1 Dose Of Study Drug (Safety Population) | 8 | 40 | 39
Dose-limiting Toxicity (DLT) Evaluable (A participant that experienced an adverse event (AE) meeting DLT criteria during Cycle 1 or who received the full dose of atezolizumab and all doses of entinostat during Cycle 1 without experiencing a DLT was considered DLT evaluable.) | 6 | 0 (DLTs were not evaluated in Phase 2.) | 0 (DLTs were not evaluated in Phase 2.)
Completed | 0 | 0 | 0
Not Completed | 8 | 40 | 41
Not completed — Withdrawal by Subject | 4 | 12 | 12
Not completed — Death | 4 | 19 | 21
Not completed — Lost to Follow-up | 0 | 3 | 3
Not completed — Study Terminated By Sponsor | 0 | 5 | 4
Not completed — Other than Specified | 0 | 0 | 1
Not completed — Discontinued Treatment but Remained in Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: all randomized participants.
Groups:
- Phase 2 Expansion: Entinostat Plus Atezolizumab: Participants received entinostat 5 mg in combination with atezolizumab 1200 mg.
- Phase 2 Expansion: Placebo Plus Atezolizumab: Participants received placebo in combination with atezolizumab 1200 mg.
- Total: Total of all reporting groups
Arm/Group | Phase 1b Dose Determination: Entinostat Plus Atezolizumab | Phase 2 Expansion: Entinostat Plus Atezolizumab | Phase 2 Expansion: Placebo Plus Atezolizumab | Total
Number analyzed (Participants) | 8 | 40 | 41 | 89
Age, Continuous [Mean (Full Range); unit: years] | 57.5 [39.0 to 75.0] | 56.9 [32.0 to 81.0] | 54.3 [29.0 to 87.0] | 56.2 [29.0 to 87.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 40 | 41 | 89
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 10 | 17
  Not Hispanic or Latino | 6 | 35 | 30 | 71
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 6 | 30 | 30 | 66
  Race: Black Or African American | 2 | 5 | 8 | 15
  Race: Asian | 0 | 3 | 0 | 3
  Race: Other | 0 | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Participants Experiencing DLT
Description: Phase 1b employed a classical 3+3 design, with the determination of DLT based on entinostat in combination with atezolizumab within the first cycle of treatment (that is, between Day 1 to Day 21 of Cycle 1). Six participants were required to be treated in a dose level for it to be considered MTD or the Recommended Phase 2 Dose (RP2D). A DLT was defined as the occurrence of specific events, defined in the protocol, that were considered by the investigator to be at least possibly related to study drug using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version 4.03.The DLT assessment window (Cycle 1) was the time period between Cycle 1 Day 1 until Cycle 2 Day 1 (expected to be 21 days after Cycle 1 Day 1).
Time Frame: Up to 21 days after Cycle 1 Day 1
Population: A participant that experienced an adverse event (AE) meeting DLT criteria during Cycle 1 or who received the full dose of atezolizumab and all doses of entinostat during Cycle 1 without experiencing a DLT was considered DLT evaluable.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1b Dose Determination: Entinostat Plus Atezolizumab: Participants received entinostat 5 mg on Days 1, 8, and 15 along with atezolizumab 1200 mg via intravenous (IV) infusion on Day 1 of Cycle 1 (21- day cycle).
Arm/Group | Phase 1b Dose Determination: Entinostat Plus Atezolizumab
Number analyzed (Participants) | 6
Participants | 0

2. Primary Outcome: Phase 1b: Determination of the RP2D
Description: Phase 1b employed a classical 3+3 design, with the determination of the RP2D based on entinostat in combination with atezolizumab within the first cycle of treatment (that is, between Day 1 to Day 21 of Cycle 1). The RP2D was defined as equal to or less than the preliminary maximum tolerated dose (MTD) and was determined in discussion with the sponsor, the study medical monitor, and dose determination phase investigators. The MTD was defined as the highest dose level at which <33% of 6 participants experience DLT.
Time Frame: Up to 21 days after Cycle 1 Day 1
Population: Participants evaluable for DLTs. A participant that experienced an AE meeting DLT criteria during Cycle 1 or who received the full dose of atezolizumab and all doses of entinostat during Cycle 1 without experiencing a DLT was considered DLT evaluable.
Measure: Number; unit: milligram
Groups:
- Phase 1b Dose Determination: Entinostat Plus Atezolizumab: Participants received entinostat 5 mg on Days 1, 8, and 15 along with atezolizumab 1200 mg via IV infusion on Day 1 of Cycle 1 (21-day cycle).
Arm/Group | Phase 1b Dose Determination: Entinostat Plus Atezolizumab
Number analyzed (Participants) | 6
milligram | 5

3. Primary Outcome: Phase 2 Expansion: Duration of Progression-free Survival (PFS) Using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: The duration of PFS, assessed using RECIST 1.1, was used to evaluate the efficacy of entinostat at the RP2D in combination with atezolizumab in participants with advanced triple negative breast cancer (aTNBC). It was defined as the number of months from randomization to the earlier of progressive disease or death due to any cause. One month was considered 30.4375 days. PFS (months) = (Date of Progression or Censoring - Date of Randomization + 1)/30.4375.
Time Frame: Up to 1 year
Population: Full Analysis Set (FAS): all participants who were randomized to study treatment, regardless of whether they actually received study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2 Expansion: Entinostat Plus Atezolizumab | Phase 2 Expansion: Placebo Plus Atezolizumab
Number analyzed (Participants) | 40 | 41
months | 1.68 [1.41 to 3.09] | 1.51 [1.41 to 2.43]

4. Secondary Outcome: Phase 2 Expansion: Duration of PFS Using Immune Response RECIST (irRECIST)
Description: The duration of PFS, assessed using irRECIST, was used to evaluate the efficacy of entinostat at the RP2D in combination with atezolizumab in participants with aTNBC. It was defined as the number of months from randomization to the earlier of progressive disease or death due to any cause. One month was considered 30.4375 days. PFS (months) = (Date of Progression or Censoring - Date of Randomization + 1)/30.4375.
Time Frame: Up to 1 year
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2 Expansion: Entinostat Plus Atezolizumab | Phase 2 Expansion: Placebo Plus Atezolizumab
Number analyzed (Participants) | 40 | 41
months | 1.68 [1.45 to 3.81] | 1.54 [1.41 to 2.83]

5. Secondary Outcome: Phase 2 Expansion: Overall Response Rate (ORR) Using RECIST 1.1 and irRECIST
Description: ORR was defined as the crude percentage of participants achieving a best overall response of complete response (CR) or partial response (PR) assessed using RECIST 1.1 and irRECIST. ORR calculated as: (number of participants with best overall response as CR or PR)/total number of participants. The overall response was determined locally by the investigator at each scheduled assessment.
Time Frame: Up to 1 year
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2 Expansion: Entinostat Plus Atezolizumab | Phase 2 Expansion: Placebo Plus Atezolizumab
Number analyzed (Participants) | 40 | 41
percentage of participants
  ORR per RECIST 1.1 | 12.5 | 2.4
  ORR per irRECIST 1.1 | 12.5 | 2.4

6. Secondary Outcome: Phase 2 Expansion: Clinical Benefit Rate (CBR) Using RECIST 1.1 and irRECIST
Description: CBR was estimated based on the crude percentage of participants in each treatment arm whose best overall response during the course of study treatment was CR, PR, or stable disease (SD) lasting for at least 24 weeks (measured from the date of randomization to the last date where SD was reported).
Time Frame: Up to 1 year
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Groups:
- Phase 2 Entinostat Plus Atezolizumab: Participants received entinostat 5 mg in combination with atezolizumab 1200 mg.
- Placebo Plus Atezolizumab: Participants received placebo in combination with atezolizumab 1200 mg.
Arm/Group | Phase 2 Entinostat Plus Atezolizumab | Placebo Plus Atezolizumab
Number analyzed (Participants) | 40 | 41
percentage of participants
  CBR per RECIST 1.1 | 15.0 | 7.3
  CBR per irRECIST 1.1 | 15.0 | 7.3

7. Secondary Outcome: Phase 2 Expansion: Overall Survival (OS)
Description: OS was defined as the number of months from randomization to date of death from any cause. Participants who were alive or lost to follow-up as of a data analysis cutoff date were right-censored. One month was considered 30.4375 days. OS (months) = (Date of Death/Censoring - Date of Randomization + 1)/30.4375
Time Frame: Up to 5 years
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2 Expansion: Entinostat Plus Atezolizumab | Phase 2 Expansion: Placebo Plus Atezolizumab
Number analyzed (Participants) | 40 | 41
months | 12.25 [5.49 to 21.16] | 11.20 [7.43 to 15.77]

8. Secondary Outcome: Phase 2 Expansion: Duration of Response (DOR)
Description: DOR was defined as the number of months from the date where a CR/PR (based on RECIST 1.1) or immune response CR (irCR)/immune response PR (irPR) was firstly observed, to the first date that recurrent or progressive disease was documented.
Time Frame: Up to 2 years
Population: Data was not collected to estimate DOR using the prespecified Kaplan-Meier method for this outcome measure.
Arm/Group | Phase 2 Expansion: Entinostat Plus Atezolizumab | Phase 2 Expansion: Placebo Plus Atezolizumab
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Phase 2 Expansion: Time To Response (TTR)
Description: TTR was defined for the subset of participants that achieved best overall response of confirmed CR/PR or confirmed irCR/irPR as the number of months from date of randomization to date of the initial documented response of CR/PR (based on RECIST 1.1) or irCR/irPR (based on irRECIST).
Time Frame: Up to 2 years
Population: Data was not collected to estimate TTR using the prespecified Kaplan-Meier method for this outcome measure.
Arm/Group | Phase 2 Expansion: Entinostat Plus Atezolizumab | Phase 2 Expansion: Placebo Plus Atezolizumab
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 5 years
Description: All-cause mortality based upon all enrolled participants (ITT population), regardless of whether treatment was received. Serious and other adverse events based upon participants that received at least 1 dose of study drug (safety population).
Groups:
- Phase 1 Dose Determination Phase: Entinostat Plus Atezolizumab; Phase 2 Expansion: Entinostat Plus Atezolizumab: Participants received entinostat 5 mg in combination with atezolizumab 1200 mg.
Arm/Group | Phase 1 Dose Determination Phase: Entinostat Plus Atezolizumab | Phase 2 Expansion: Entinostat Plus Atezolizumab | Phase 2 Expansion: Placebo Plus Atezolizumab
All-Cause Mortality (participants affected / at risk) | 4/8 | 20/40 | 21/41
Serious Adverse Events (participants affected / at risk) | 2/8 | 18/40 | 14/39
Other Adverse Events (participants affected / at risk) | 8/8 | 34/40 | 30/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 Dose Determination Phase: Entinostat Plus Atezolizumab (N=8) | Phase 2 Expansion: Entinostat Plus Atezolizumab (N=40) | Phase 2 Expansion: Placebo Plus Atezolizumab (N=39)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Cardiac Arrest (Cardiac disorders) | 0 | 1 | 0
Cardiac Tamponade (Cardiac disorders) | 0 | 0 | 1
Cardiopulmonary Failure (Cardiac disorders) | 0 | 1 | 0
Pericardial Effusion (Cardiac disorders) | 0 | 0 | 2
Sinus Tachycardia (Cardiac disorders) | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Gait Disturbance (General disorders) | 0 | 1 | 0
Oedema Peripheral (General disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 2 | 1
Biliary Obstruction (Hepatobiliary disorders) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 2 | 0
Infectious Mononucleosis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0
Blood Bilirubin Increased (Investigations) | 0 | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Brain Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Spinal Cord Compression (Nervous system disorders) | 1 | 0 | 0
Mental Status Changes (Psychiatric disorders) | 0 | 0 | 2
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 2
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0
Pelvic Venous Thrombosis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 Dose Determination Phase: Entinostat Plus Atezolizumab (N=8) | Phase 2 Expansion: Entinostat Plus Atezolizumab (N=40) | Phase 2 Expansion: Placebo Plus Atezolizumab (N=39)
Anaemia (Blood and lymphatic system disorders) | 0 | 8 | 5
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 6 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 9 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 3
Vision Blurred (Eye disorders) | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 6 | 2
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 7 | 6
Constipation (Gastrointestinal disorders) | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 13 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 0
Eructation (Gastrointestinal disorders) | 1 | 0 | 0
Indigestion (Gastrointestinal disorders) | 0 | 2 | 2
Loose Stool (Gastrointestinal disorders) | 0 | 5 | 0
Nausea (Gastrointestinal disorders) | 0 | 14 | 4
Nausea (Gastrointestinal disorders) | 5 | 0 | 0
Nausea (Intermittent) (Gastrointestinal disorders) | 0 | 0 | 2
Stomach Cramping (Gastrointestinal disorders) | 0 | 3 | 0
Vomiting (Gastrointestinal disorders) | 0 | 9 | 5
Vomiting (Intermittent) (Gastrointestinal disorders) | 0 | 1 | 2
Chills (General disorders) | 0 | 3 | 3
Fatigue (General disorders) | 0 | 25 | 14
Fatigue (General disorders) | 6 | 0 | 0
Fever (General disorders) | 0 | 8 | 7
Flu Like Symptoms (General disorders) | 0 | 0 | 2
Lack of Energy (General disorders) | 0 | 2 | 2
Oedema (General disorders) | 1 | 0 | 0
Oedema Peripheral (General disorders) | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 0
Weakness (General disorders) | 0 | 2 | 2
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 3 | 2
Urinary Tract Infection (Infections and infestations) | 0 | 3 | 1
Urinary Tract Infection (Infections and infestations) | 2 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 2
Alanine Aminotransferase Increased (Investigations) | 0 | 3 | 1
Alkaline Phosphatase Increased (Investigations) | 0 | 4 | 0
Decreased White Blood Count (Investigations) | 0 | 3 | 0
Increased Creatinine (Investigations) | 0 | 1 | 2
Neutrophil Count Decreased (Investigations) | 0 | 3 | 2
Platelet Count Decreased (Investigations) | 0 | 7 | 0
Weight Decreased (Investigations) | 1 | 0 | 0
Weight Loss (Investigations) | 0 | 4 | 2
White Blood Cell Count Decreased (Investigations) | 0 | 3 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 3 | 3
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1 | 3
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 4 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 4 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 4 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Loss of Appetite (Metabolism and nutrition disorders) | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Limb Mass (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Right Hip Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Right Leg Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 4 | 3
Dizziness (Nervous system disorders) | 2 | 0 | 0
Dygeusia (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 9 | 7
Intermittent Headache (Nervous system disorders) | 0 | 3 | 1
Taste Disturbance (Nervous system disorders) | 0 | 0 | 2
Depressed Mood (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 3 | 7
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Breast Pain (Reproductive system and breast disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Dry Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 2
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema Nodosum (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 4 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin Burning Sensation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hot Flashes (Vascular disorders) | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of the results of the multi-center Study shall not be made before the first multi-site publication by Sponsor or Publications Committee. No Public Presentation by Institution or Investigator will be made until Study Documentation/Results from all sites are received and analyzed by Sponsor. Separate publication by Investigator will be delayed for a period of 18 months until the initial publication by Committee or Sponsor, or a determination is made not to make such publication.

DOCUMENTS (2):
  • Study Protocol (2018-09-11): https://cdn.clinicaltrials.gov/large-docs/80/NCT02708680/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-08): https://cdn.clinicaltrials.gov/large-docs/80/NCT02708680/SAP_001.pdf